CLINICAL TRIAL: NCT03475719
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristic After Administration of Fixed-dose Combination or Loose Combination of HUG186 in Healthy Adult Male or Menopausal Female Volunteers
Brief Title: A Clinical Trial to Evaluate the Safety and Pharmacokinetic
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUG186_P1
Record Dates: First submitted 2018-01-11; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, single-dose, two-treatment, two-sequence, two-way crossover study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUG186-B and HUG186-D (Active Comparator): Bazedoxifene acetate 22.6mg, Cholecalciferol 8.0mg(=800IU)
  Interventions: Drug: HUG186-B and HUG186-D
- HUG186 (Experimental): Combination of Bazedoxifene acetate 22.6mg and Cholecalciferol 8.0mg(=800IU)
  Interventions: Drug: HUG186

INTERVENTIONS:
Drug: HUG186-B and HUG186-D — Bazedoxifene acetate 22.6mg, Cholecalciferol 8.0mg(=800IU)
  Arms: HUG186-B and HUG186-D
Drug: HUG186 — Combination of Bazedoxifene acetate 22.6mg and Cholecalciferol 8.0mg(=800IU)
  Arms: HUG186

SUMMARY:
A phase 1 clinical trail to evaluate the safety and pharmacokinetic characteristic after administration of fixed-dose combination or loose combination of HUG186 in healthy adult male or menopausal female volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Men, age≥19 years of age, Postmenopausal women are eligible. Postmenopausal is defined as any of the following:

   * Amenorrhea for 12 or more months
   * FSH and estradiol in the postmenopausal range per local normal range.
2. Body weight of ≥ 55 kg, BMI 18.5 to 30.0
3. No morbid symptom or sign, based on physical examination, with no innate or chronic disease.
4. Subject that is considered appropriate for participating in the study by an investigator, based on clinical laboratory test (hematology, clinical chemistry, urinalysis) that is performed according to the characteristics of investigational drugs.
5. Subject that agree to apply sun cream in case of daylight exposure for more than 1hours
6. Subjects must be able to listen to and understand the detailed statement of informed consent, and willing to decide to participate in the study, follow the study directions and provide written informed consent.

Exclusion Criteria:

1. A clinically significant disease or history in hepatobiliary system, kidney, digestive system, respiratory system, hemato-oncological system, endocrine system, neuro-psychiatric system, musculo-skeletal system, immune system, otorhinolaryngological system or cardiovascular system.
2. A history of hypersensitivity to investigational drugs and its additives or clinically significant hypersensitivity to any other drug.
3. History of drug abuse, or positive in drug screening test.
4. Use of inducer or inhibitor of metabolic enzymes for drugs like barbiturate.
5. Use of any prescribed drugs or herbal remedies within 2 weeks, or use of any over-the-counter medication within 1 week prior to the first administration of investigational drug, and this will affect this study or the safety of the subjects at discretion of study investigator.
6. Participation in another clinical trial or a bioequivalent study within 3 months prior to the first administration of investigational drug (The finish time of previous study is the day of the last administration of study drug)
7. Whole blood donation within 2 months or component donation within 1 month, prior to the first administration of investigational drug, or transfusion within 1 month prior to the first administration of investigational drug.
8. Prolonged excessive alcohol consumption (>21 units/week, 1 unit=10g of pure alcohol), or subjects who can not abstain from drinking from 24 hours prior to hospitalization until the discharge.
9. Smoking more than 10 cigarettes per day, excessive caffeine consumption (example: instant coffee > 5 cups/day)
10. Subjects who are judged to be inappropriate for this study by investigators according to other reasons including clinical lab test result

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-t of Bazedoxifene | 0, 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h(17points)
  Area under the curve(AUCt) of Bazedoxifene
Cmax of Bazedoxifene | 0, 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h(17points)
  Maximum observed concentration(Cmax) of Bazedoxifene
AUC0-t of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h(18points)
  Area under the curve(AUCt) of Cholecalciferol
Cmax of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h(18points)
  Maximum observed concentration(Cmax) of Cholecalciferol

SECONDARY OUTCOMES:
Tmax of Bazedoxifene | 0, 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h(17points)
  Tmax of Bazedoxifene
AUCinf of Bazedoxifene | 0, 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h(17points)
  AUCinf of Bazedoxifene
t1/2 of Bazedoxifene | 0, 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h(17points)
  t1/2 of Bazedoxifene
Tmax of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h(18points)
  Tmax of Cholecalciferol
AUCinf of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h(18points)
  AUCinf of Cholecalciferol
t1/2 of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h(18points)
  t1/2 of Cholecalciferol

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Gyeonggi-do, Seongnam-si, South Korea